CLINICAL TRIAL: NCT02921269
Title: A Phase 2 Study of Atezolizumab (MPDL3280A) in Combination With Bevacizumab in Patients With Recurrent, Persistent or Metastatic Cervical Cancer
Brief Title: Atezolizumab and Bevacizumab in Treating Patients With Recurrent, Persistent, or Metastatic Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01430; NCI-2016-01430 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-183; 10010 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10010 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Recurrent Cervical Carcinoma; Stage IV Cervical Cancer AJCC v6 and v7; Stage IVA Cervical Cancer AJCC v6 and v7; Stage IVB Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab, bevacizumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Biological: Bevacizumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well atezolizumab and bevacizumab work in treating patients with cervical cancer that has come back, remains despite treatment, or has spread to other places in the body. Monoclonal antibodies, such as atezolizumab and bevacizumab, may shrink tumor cell and interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the anti-tumor activity (proportion of patients with objective response by Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1] criteria) of atezolizumab and bevacizumab in patients with recurrent, persistent or metastatic cervical cancer.

SECONDARY OBJECTIVES:

I. To estimate the duration of progression free survival (PFS) and overall survival (OS).

II. To assess safety by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v.5.0).

III. To describe the efficacy of the combination of atezolizumab and bevacizumab as measured by objective response, by PD-L1 expression on tumor and immune cells measured by semi-quantitative immunohistochemistry (IHC).

IV. To describe the efficacy of the combination of atezolizumab and bevacizumab as measured by objective response, by intratumoral and peripheral T-cell receptor (TCR) clonality and tumor infiltrating lymphocyte proportion.

OUTLINE:

Patients receive atezolizumab intravenously (IV) over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease per RECIST 1.1; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam; to be considered pathologically enlarged and measurable, a lymph node must be >= 15 mm (>= 1.5 cm) in short axis
* Patients must have had one prior systemic chemotherapeutic regimen for management of recurrent, persistent or metastatic carcinoma of the cervix (e.g.; paclitaxel/cisplatin, paclitaxel/cisplatin/bevacizumab), at least one which must have contained bevacizumab

  * NOTE: Patients are allowed to receive 1-2 prior regimens for management of recurrent, persistent or metastatic carcinoma of the cervix; patients who have received more than two prior systemic regimens for management of recurrent, persistent or metastatic carcinoma of the cervix are NOT eligible
  * NOTE: Prior adjuvant therapy is NOT counted as a systemic chemotherapeutic regimen for management of recurrent, persistent or metastatic carcinoma of the cervix; adjuvant therapy includes cisplatin given concurrent with primary radiation therapy (CCRT) and adjuvant chemotherapy given following the completion of concurrent chemotherapy and radiation therapy (e.g., paclitaxel and carboplatin for up to 4 cycles)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Creatinine =< 1.5 x ULN
* International normalized ratio (INR) and activated partial thromboplastin time aPTT =< 1.5 x ULN (This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* Urine protein must be screened by urinalysis; if protein is 2+ or higher, 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment
* Patient must have recurrent, persistent or metastatic cervical cancer including squamous cell, adenocarcinoma and adenosquamous histologies; mesonephric carcinoma, minimal deviation/adenoma malignum, clear cell carcinoma and gastric type are excluded
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of atezolizumab; fertile women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of bevacizumab therapy; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Tumors within previous radiated field will be designated "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Willingness to undergo a tumor biopsy

Exclusion Criteria:

* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (other than alopecia) due to agents administered more than 4 weeks earlier; however, the following therapies are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to cycle 1, day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to cycle 1, day 1)
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Prior treatment with anti-CTLA-4 therapeutic antibody or pathway-targeting agents
* Treatment with any other investigational agent within 4 weeks prior to cycle 1, day 1
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia; use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Patients with known brain metastases should be excluded from this clinical trial
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab or atezolizumab
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to cycle 1, day 1; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with atezolizumab and/or bevacizumab
* Malignancies other than the cervical cancer within 5 years prior to cycle 1, day 1, with the exception of those with a negligible risk of metastasis or death, such as adequately controlled basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the breast
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1
* Patients with clinically significant cardiovascular disease are excluded

  * Inadequately controlled hypertension (HTN) (systolic blood pressure [SBP] >= 160 mmHg and/or diastolic blood pressure [DBP] >= 90 mmHg despite antihypertensive medication)
  * History of cerebrovascular accident (CVA) within 6 months
  * Myocardial infarction or unstable angina within 6 months
  * New York Heart Association class II or greater congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* History of abdominal/pelvic fistula, gastrointestinal perforation and/or intraabdominal abscess within 6 months prior to day 1
* Evidence of bleeding diathesis or clinically significant coagulopathy
* Serious or non-healing wound, active ulcer or bone fracture
* Patients requiring treatment with a RANKL inhibitor (e.g. denosumab) who cannot discontinue it before treatment with atezolizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire F Friedman, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (22):
- United States (22):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of Colorado Hospital, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Friedman CF, Snyder Charen A, Zhou Q, Carducci MA, Buckley De Meritens A, Corr BR, Fu S, Hollmann TJ, Iasonos A, Konner JA, Konstantinopoulos PA, Modesitt SC, Sharon E, Aghajanian C, Zamarin D. Phase II study of atezolizumab in combination with bevacizumab in patients with advanced cervical cancer. J Immunother Cancer. 2020 Oct;8(2):e001126. doi: 10.1136/jitc-2020-001126. PMID 33004542

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Started | 11
Completed | 10
Not Completed | 1
Not completed — Did not complete DLT period | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 48 [31 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Rate (ORR, Either Partial or Complete Response) Defined by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Criteria
Description: Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, Complete Response (CR) is the disappearance of all lesions and Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Overall Response (OR) is CR+PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 11
Participants | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study and an absolute increase of at least 5 mm (0.5 cm) or the appearance of one or more new lesions.
Time Frame: From start of treatment to investigator determined date of progression, or death due to any cause, whichever occurs first, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 11
months | 2.9 [1.8 to 6]

3. Secondary Outcome: Overall Survival (OS)
Description: The duration of OS will be estimated.
Time Frame: From start of treatment to death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 11
months | 8.9 [3.4 to 21.9]

4. Secondary Outcome: Percent of Participants With Adverse Events
Description: The frequency and severity of adverse events will be assessed in those patients who initiate their study treatment.
Time Frame: Up to 30 days after the last dose of study treatment, on average of 4 months
Population: Overall rate of grade 3-4 adverse events attributable to study drug.
Measure: Number; unit: percent of participants
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 11
percent of participants | 36.4

5. Secondary Outcome: PD-L1 Expression on Tumor and Immune Cells Measured by Semi-quantitative Immunohistochemistry
Description: The efficacy of the combination of atezolizumab and bevacizumab as measured by objective response, will be described in patients according to PD-L1 positive and PD-L1 negative.
Time Frame: Up to 2 years
Population: The 8 participants with adequate pretreatment core biopsies were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 8
Participants | 3

6. Secondary Outcome: Intratumoral and Peripheral T-cell Receptor (TCR) Clonality Assessed by TCR Sequencing
Description: Will be used to describe the efficacy of the combination of atezolizumab and bevacizumab.
Time Frame: Up to 2 years
Population: The 8 participants with adequate pretreatment core biopsies were included in the analysis. However, there were insufficient samples to run this assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 8
Participants | 0

7. Other Pre Specified Outcome: Tumor Infiltrating Lymphocyte Proportion
Description: Will be used to describe the efficacy of the combination of atezolizumab and bevacizumab.
Time Frame: Up to 2 years
Population: The 8 participants with adequate pretreatment core biopsies were included in the analysis.
Measure: Median (Full Range); unit: percent of CD8 in the tumor
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
Number analyzed (Participants) | 8
percent of CD8 in the tumor | 1.17 [0.06 to 2.77]

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study treatment, on average of 4 months.
Arm/Group | Treatment (Atezolizumab, Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 11/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Atezolizumab, Bevacizumab) (N=11)
Sinus tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Stroke (Cardiac disorders) | 1
Thromboembolic event (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Gastrointestinal disorders) | 2
Lipase increased (Gastrointestinal disorders) | 1
Alkaline phosphatase increased (Gastrointestinal disorders) | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 2
Gastrointestinal bleeding (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Fever (General disorders) | 3
Pain (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalagia (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Arachnoiditis (Nervous system disorders) | 1
Sensorineural hearing loss (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Depression (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Meningitis (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT02921269/Prot_SAP_000.pdf